CLINICAL TRIAL: NCT02063386
Title: A Phase I, Single-centre, Open-label Study to Assess the Absorption, Distribution, Metabolism and Excretion (ADME) of a Single Oral Dose of 14C-labelled AZD1722 in Healthy Male Volunteers
Brief Title: AZD1722 Open Label, Absorption Distribution Metabolism and Excretion Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5611C00007
Record Dates: First submitted 2014-02-13; First posted 2014-02-14 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1722 (Experimental): Single oral dose 15 mg of [14C]AZD1722
  Interventions: Drug: AZD1722

INTERVENTIONS:
Drug: AZD1722 — Single oral dose 15 mg of [14C]AZD1722

SUMMARY:
To assess the absorption, distribution, metabolism and excretion of a single dose of 14C labelled AZD1722 in order to define the rates and routes of elimination of AZD1722 and if formed, metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged ≥50 years
* Regular daily bowel movements.
* Have a body mass index (BMI) between 18 and 32 kg/m2 (inclusive) and weigh at least 50 kg and no more than 110 kg.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of GI, hepatic or renal disease including GI surgery other than appendectomy or any other condition known to interfere with the ADME of drugs.
* Loose stools (Bristol Stool Form Score of 6 or 7) ≥2 days in the past 7 days before admission to the study centre
* Use of medications that are known to affect stool consistency and/or GI motility, including fibre supplements, anti-diarrheals, prokinetic drugs, enemas, probiotic medications or supplements; or salt or electrolyte supplements containing sodium, potassium, chloride, or bicarbonate formulations during the past 7 days before admission to the study centre.
* Volunteers exposed to radiation levels above background (eg, via X-ray examination) of >5 mSv in the last year, >10 mSv over the last 5 years or a cumulative total of >1 mSv per year of life.
* Participation in a previously radiolabelled study within the last 5 years

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and feces | Day 1: Pre-dose and up to 168 hours post-dose
Total percentage of radioactive dose recovered from both urine and feces | Day 1: Pre-dose and up to 168 hours post-dose
Concentration of total radioactivity in blood and plasma samples | Timeframe: Day 1: Predose and up to 120 hours
Concentration of AZD1722 in plasma samples | Timeframe: Day 1: Predose and up to 120 hours

SECONDARY OUTCOMES:
Safety variables (adverse events, vital signs, ECGs, clinical laboratory tests) | up to 50 days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2458&filename=d5611c00007-study-synopsis_Redacted.pdf